CLINICAL TRIAL: NCT02653131
Title: The Use of Dipeptidyl Peptidase-4 Inhibitor Influences the Absorption of Intestine in Short Bowel Syndrome
Brief Title: The Use of DPP-4 Inhibitors in Short Bowel Syndrome
Acronym: DPP-4
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: too many side-effects
Sponsor: Stanley Dudrick's Memorial Hospital (Other)
Responsible Party: Principal Investigator, Stanislaw Klek, Assoc. Prof., Stanley Dudrick's Memorial Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLP-1
Record Dates: First submitted 2016-01-10; First posted 2016-01-12 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Short Bowel Syndrome
Keywords: Short bowel syndrome
MeSH Terms: conditions — Short Bowel Syndrome | interventions — Dipeptidyl-Peptidase IV Inhibitors; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DPP-4 (Experimental): The administration of the DPP-4 inhibitor in the form of a pill once per day
  Interventions: Drug: Dipeptidyl peptidase-4 inhibitor
- NO DPP (No Intervention): no therapy

INTERVENTIONS:
Drug: Dipeptidyl peptidase-4 inhibitor
  Other Names: Sitagliptin
  Arms: DPP-4

SUMMARY:
The inhibition of Dipeptidyl peptidase-4 should increase the concentration of glucagone-like peptide 1 and 2, and the increase of the latter should increase the absorptive capacity of the intestine.

DETAILED DESCRIPTION:
The only effective (to some extend drug) in short bowel syndrome is Glucacone-like peptide 4. Its price is, however, to high to really change the treatment strategy for intestinal failure. The Dipeptidyl peptidase-4 inhibitor, which a drug which is commonly used in the treatment of diabetes mellitus type II, should increase the concentration of glucagone-like peptide 1 and 2, and the increase of the latter should increase the absorptive capacity of the intestine.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving home parenteral nutrition (HPN) because of short bowel syndrome for at least 12 months
* stable metabolic status
* benign disease

Exclusion Criteria:

* HPN < 12 months
* metabolically unstable
* cancer as the reason for intestinal failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-01; Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Improvement of intestinal absorption | 12 months
  the use of DPP-4 inhibitor results in the better intestinal absorption

CONTACTS AND LOCATIONS:
Locations (1):
- Stanley Dudrick's Memorial Hospital, Skawina, Poland

IPD SHARING:
Plan to Share IPD: No
All data is a part of a research

REFERENCES:
- [Background] Jeppesen PB. Pharmacologic options for intestinal rehabilitation in patients with short bowel syndrome. JPEN J Parenter Enteral Nutr. 2014 May;38(1 Suppl):45S-52S. doi: 10.1177/0148607114526241. Epub 2014 Mar 10. PMID 24615689